CLINICAL TRIAL: NCT01668901
Title: A Randomized Controlled Prospective Trial of Warfarin Versus Aspirin for Stroke Prevention in Patients With Atrial Fibrillation and Chronic Kidney Disease
Brief Title: Warfarin Versus Aspirin in Patients With Atrial Fibrillation and Chronic Kidney Disease
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Financial problem
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WASAK
Record Dates: First submitted 2012-08-16; First posted 2012-08-20 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2012-08

CONDITIONS: Atrial Fibrillation; Chronic Kidney Disease
Keywords: warfarin; aspirin
MeSH Terms: conditions — Atrial Fibrillation; Renal Insufficiency, Chronic | interventions — Warfarin; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- warfarin (Experimental): medication
  Interventions: Drug: warfarin
- aspirin (Active Comparator): medication
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: warfarin — anticoagulation
  Arms: warfarin
Drug: Aspirin — antiplatelet
  Arms: aspirin

SUMMARY:
In this study, the investigators examine whether aspirin or warfarin is useful for atrial fibrillation patients with chronic kidney disease.

DETAILED DESCRIPTION:
randomised open labelled prospective study

We enroll patients with CHADS2 score 1 non-valvular AF with chronic kidney disease, and analyze all thromboembolic event or major bleeding event during follow-up period. Warfarin group take dose adjusted warfarin (target INR 2.0-3.0) and aspirin group take aspirin 100mg daly.

Thromboembolic events: Ischemic stroke or systemic arterial occlusion Major bleeding: gastrointestinal bleeding or intracranial bleeding (code 430, code 431, code 432 by ICD-9-CM codes)

-> Only the first event of each case will be used for the analysis

ELIGIBILITY:
Inclusion Criteria:

* CHADS2 score 1 nonvalvular atrial fibrillation patients with chronic kidney disease

Exclusion Criteria:

* HAS-BLED ≥30
* History of syncope or seizure within 1 year
* History of major bleeding event within 6 months
* BP>180/100
* Abnormal prothrombin time
* Hypersensitivity of aspirin or warfarin
* Folstein mini mental state examination score <26
* Taking or had taken other anticoagulants

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2015-09 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Thromboembolic event | through study completion, an average of 1 year
  Ischemis stroke and systemic thromboembolism

SECONDARY OUTCOMES:
Major bleeding | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Seil Oh, MD,PhD, Principal Investigator — Seoul National University Hospital, Seoul , Korea
Locations (1):
- Seoul Nationap University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No